CLINICAL TRIAL: NCT02197013
Title: Evaluation of Introcan Safety 3 Closed IV Catheter
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HC-O-H-1207
Record Dates: First submitted 2014-07-17; First posted 2014-07-22 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Patients in Need for Intravenous Access

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Introcan Safety 3: Closed IV Catheter
- Introcan Safety: IV catheter

SUMMARY:
Incidence and time of occurrence of blood leakage with the closed intravascular catheter Introcan Safety 3 in comparison to Introcan Safety

ELIGIBILITY:
Inclusion Criteria:

* need for intravenous access

Exclusion Criteria:

* n. a.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in need for intravenous access
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Frequency and time of occurence of blood leakage | Within one minute

SECONDARY OUTCOMES:
Problems during catheter insertion and fixation of Introcan Safety 3 | During insertion and fixation of catheter
Necessity of disconnection of catheter | During catheter placement

CONTACTS AND LOCATIONS:
Overall Officials: Gertrud Haeseler, Prof., Principal Investigator — KKRN
Locations (1):
- KKRN Katholisches Klinikum Ruhrgebiet Nord GmbH (KKRN), Dorsten, Germany